CLINICAL TRIAL: NCT02824250
Title: Mindfulness and Migraine: A Randomized Controlled Trial
Brief Title: Mindfulness and Migraine Research Study
Acronym: M&M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Kaiser Permanente (Other); Sutter Health (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 897613; 1R01AT00908101 (Other Grant/Funding Number: National Center for Complementary and Integrative Health)
Record Dates: First submitted 2016-06-07; First posted 2016-07-06 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Migraine; Chronic Pain
Keywords: Migraine; Mindfulness; MBSR
MeSH Terms: conditions — Migraine Disorders; Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR + Usual Care (Experimental): 8-week standard Mindfulness-Based Stress Reduction (MBSR) course + standard of care
  Interventions: Behavioral: MBSR
- Usual Care (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: MBSR — Mindfulness-Based Stress Reduction (MBSR) is an 8-week classroom based program of mindfulness meditation and gentle yoga.
  Arms: MBSR + Usual Care

SUMMARY:
The primary aim of this study is to conduct a randomized controlled feasibility trial of MBSR for patients with moderate-to- severe migraine headache.

DETAILED DESCRIPTION:
Migraine, one of the most common neurological disorders in the U.S., is ranked among the top 20 causes of disability worldwide. Migraine is currently one of the leading causes of disease burden for women aged 15-44 years and affects an estimated 11% of the adult population globally, with a strong female predominance. Current approaches to therapy are primarily medication-based but are limited by often-inadequate effectiveness, high costs for many migraine-specific medications, and common side effects. In addition, there likely exist subtypes of migraine that may affect the likelihood of response to treatment, but these have been poorly investigated to-date. Furthermore, many patients are interested in exploring alternatives to pharmacological therapy for this functional disorder.

Mindfulness-based stress reduction (MBSR), a meditation-based intervention developed by Kabat-Zinn at the University of Massachusetts, has been increasingly shown to be effective for many patients with a variety of functional disorders. Recent small pilot studies suggest that MBSR may also provide an important benefit as an adjunctive therapy for patients with migraine headaches.

In preparation for a fully powered randomized controlled clinical trial of MBSR for patients with moderate-to-severe migraine headache, the investigators propose a detailed pilot/feasibility study to develop and test the clinical research methods required for a successful Phase III trial. The investigators will first identify a large number of migraineurs in the Northern California-based Sutter Health system using analytic tools previously developed by the group. Next, using latent class analysis, the investigators will identify subgroups of migraine patients defined by comorbidities. The investigators will then enroll 60 patients with a pattern of 4-20 headaches per month and randomize them to a full 8-week MBSR intervention with usual care or usual care alone, with follow-up at 4 months. The primary clinical outcome is change in headache frequency at 4 months, with several secondary outcomes, including assessments of pain, quality of life, and functional status.

As a feasibility study, the primary emphases of the trial are to demonstrate the investigators' ability to recruit and retain participants, to test whether their proposed enrollment criteria identify the appropriate patient population, to assess participants' levels of adherence to all aspects of the protocol, and to determine optimal methods for data collection. No tests of clinical effectiveness will be performed.

The results of this feasibility study will provide invaluable information for the study investigators in development of methods to ensure a highly successful and informative Phase III trial of a promising MBSR intervention for this common and distressing medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* 4-20 headaches per month (based on run-in headache diary)

Exclusion Criteria:

* No meditation or MBSR during the past 6 months
* Cognitively or emotionally impaired as judged by a research physician prior to randomization
* Pregnant
* Lack of English language skills
* No new migraine medication in past month
* Incomplete headache diary during run-in period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
recruitment rate | 18 months post recruitment start
  number recruited per month

SECONDARY OUTCOMES:
treatment adherence | 18 months post recruitment start
  proportion of classes attended
diary completion | 2 years post recruitment start
  proportion of days completed for each diary type

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto Medical Foundation Research Institute, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pressman A, Law H, Stahl R, Scott A, Jacobson A, Dean L, Sudat S, Obillo A, Avins A. Conducting a pilot randomized controlled trial of community-based mindfulness-based stress reduction versus usual care for moderate-to-severe migraine: protocol for the Mindfulness and Migraine Study (M&M). Trials. 2019 May 6;20(1):257. doi: 10.1186/s13063-019-3355-y. PMID 31060619